CLINICAL TRIAL: NCT05206955
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy of Tadalafil Versus Placebo in Improving Hemodynamics and End-Organ Dysfunction in Fontan Physiology (TRIUMPH Trial)
Brief Title: Study of Tadalafil vs. Placebo for Improving Hemodynamics and End-Organ Dysfunction in Fontan Physiology
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexander C. Egbe, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-009890; R01HL160761-01 (NIH)
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Fontan Palliation
MeSH Terms: interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tadalafil Group (Experimental): Study participants will receive 10 mg of Tadalafil daily for 1 week, then 20 mg daily for 1 week, and finally 40 mg daily for 50 weeks for a total therapy time of 52 weeks. Tadalafil will be taken orally in capsule form once daily.
  Interventions: Drug: Tadalafil
- Placebo Group (Placebo Comparator): Study participants will receive a placebo capsule that looks identical to the Tadalafil capsule. The placebo will be taken orally once daily for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — 10 mg once daily orally week 1, 20 mg once daily orally during week 2, and 40 mg once daily orally during weeks 3 through 52
  Arms: Tadalafil Group
Drug: Placebo — Looks exactly like the study drug, but it contains no active ingredient
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to find out more about the effectiveness of Tadalafil in improving hemodynamic capabilities, endothelial function, and end-organ function in patients who have previously undergone a Fontan Palliation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old.
* Have previously undergone a Fontan Palliation.
* Able to exercise using a supine bike.
* Ability and willingness to provide written consent.
* Undergoing a clinically indicated Cardiac Catheterization

Exclusion Criteria:

* Patients < 18 years old.
* Current intravenous inotropic drugs.
* Current use of alpha-blockers, pulmonary vasodilators, or nitrates.
* Unable to exercise.
* Pregnancy or lactating.
* Unable or unwilling to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Microvascular endothelial function | 52 weeks
  Measured by the reactive hyperemic index using peripheral artery tonometry (EndoPAT)
Pulmonary vascular reserve | 52 weeks
  The slope of mean pulmonary artery pressure / cardiac output (mPAP/CO)

SECONDARY OUTCOMES:
Liver stiffness | 52 weeks
  Liver magnetic resonance elastography (MRE) will be used to assess liver stiffness expressed in Pascals (Pa)
Renal function | 52 weeks
  Measured by the glomerular filtration rate
Exercise capacity | 52 weeks
  Assessed using peak VO2 (oxygen consumption) obtained from an upright treadmill or supine bike cardiopulmonary exercise test with echocardiogram
Patient reported quality of life | 52 weeks
  Measured by the Minnesota Living with Heart Failure Questionnaire that asks subjects to rate how much their heart failure (heart condition) has affected their life during the past month (4 weeks) on a scale of 0=no and 5=very much.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Egbe, MBBS, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No